CLINICAL TRIAL: NCT00213369
Title: Neuromodulation of Aspiration Secondary to Stroke
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2004/08/HP
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-02-16 (Estimated); Status verified 2012-02

CONDITIONS: Deglutition Disorders
Keywords: aspiration; stroke; motor evoked potential; cortical evoked potential; neuromodulation
MeSH Terms: conditions — Deglutition Disorders; Stroke

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Aspiration could induce major respiratory affection. They are often present after stroke. The aim of this study is to facilitate swallowing recuperation in stroke patients using peripheral laryngeal stimulation and to understand its mechanisms using motor evoked potential and cortical evoked potential.

ELIGIBILITY:
Inclusion Criteria:

stroke aspiration

Exclusion Criteria:

pace maker tracheostomy epilepsy pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: stroke patients
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2007-01; Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: eric verin, MD PHD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France